CLINICAL TRIAL: NCT05852223
Title: Neoadjuvant Pembrolizumab in High-risk Thyroid Cancers
Brief Title: Pembrolizumab in High-risk Thyroid Cancer
Acronym: NePenThe
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Laura Deborah Locati, MD, PhD, Istituti Clinici Scientifici Maugeri SpA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NePenThe; 2021-003524-32 (EudraCT Number)
Record Dates: First submitted 2023-04-26; First posted 2023-05-10 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Differentiated Thyroid Cancer
Keywords: differentiated thyroid carcinoma; neoadjuvant treatment; pembrolizumab
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- experimental arm A (Experimental): N° 20 patients: patients will receive pembrolizumab 200 mg Every Three Weeks (Q3W) for 2 courses, followed by thyroidectomy +/- radioiodine according to the risk class
  Interventions: Drug: Pembrolizumab
- control group B (No Intervention): N° 5 patients: patients will be treated for clinical practice with upfront thyroidectomy followed by +/- radioiodine according to the risk class

INTERVENTIONS:
Drug: Pembrolizumab — Neoadjuvant pembrolizumab 200mg Q3W will be administered via IV infusion for 2 courses from the date of randomization until to the date of thyroidectomy.
  Arms: experimental arm A

SUMMARY:
This window of opportunity trial is studying a checkpoint inhibitor agent to treat differentiated thyroid cancer in a neoadjuvant setting. A checkpoint inhibitor is a compound aimed at restoring tumor immunosurveillance. The name of this agent is pembrolizumab.

DETAILED DESCRIPTION:
This is a window of opportunity trial. The window of opportunity trial investigates the metabolic and/or the pharmacodynamic effect of a compound, exploiting the window of time between the diagnosis and the start of treatment, e.g surgical intervention. Pembrolizumab has been approved by FDA and EMA for several type of cancers. Pembrolizumab has not been approved for treatment against thyroid cancers. Pembrolizumab is a checkpoint inhibitor, it binds the protein PD-1 on the surface on immune cells (T cells) interrupting the cross talk with its ligands, PD-L1 and PD-L2, on cancer cells, allowing the immune system to recognize and destroy the cancer cells.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of differentiated thyroid carcinoma candidate to surgery not previously treated will be enrolled in this study.
2. Patients with a risk > 20% for persistent/recurrent disease: primary tumor > 4 cm; multifocal papillary microcarcinoma with extra tumor extension (ETE) and known BRAF V600E mutation; clinical N1; gross ETE (macroscopic invasion of perithyroidal soft tissues); extranodal extension; expected incomplete tumour resection.
3. Poorly differentiated carcinoma; Hurtle cell carcinoma.
4. Patients with distant metastasis at diagnosis.
5. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
6. Have measurable disease based on RECIST 1.1.
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of allocation/randomization.
8. Have adequate organ function as defined in the following table (Table 2) Specimens must be collected within 10 days prior to the start of study treatment.
9. Male participants:

   A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 6 months (e.g. 5 terminal half-lives for pembrolizumab) after the last dose of study treatment and refrain from donating sperm during this period.
10. female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP).
    2. a WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 4 months after the last dose of study treatment

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to randomization. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to randomization.
4. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed. Administration of killed vaccines is allowed.
6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in-situ (eg, breast carcinoma or cervical cancer in situ that have undergone potentially curative therapy are not excluded).
9. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
12. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
13. Has an active infection requiring systemic therapy.
14. History of Human Immunodeficiency Virus (HIV) infection.
15. History of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
16. Has a known history of active TB (Bacillus Tuberculosis).
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
20. Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To investigate the behavior of exhausted cytotoxic T cell (CD8+ T) in tumor tissue in response to pembrolizumab | Up to 12 months after surgery
  Relative proportion of exhausted CD8+ T cells and their topological relationships to cell clusters in TCs following neoadjuvant pembrolizumab assessed by "Spatial-transcriptomic" sequencing
To investigate the behavior of exhausted cytotoxic T cell (CD8+ T) at circulating level in response to pembrolizumab | Up to 12 months after surgery
  Relative proportion of exhausted CD8+ T cells and their topological relationships to cell clusters in TCs following neoadjuvant pembrolizumab assessed by single-cell sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Laura D Locati, MD, PhD, Principal Investigator — Istituti Clinici Scientifici Maugeri
Locations (1):
- Istituti Clinici Scientifici Maugeri, Pavia, Lombardy, Italy